CLINICAL TRIAL: NCT05341830
Title: The Effect of Recovery Housing on Patients' Health, Housing, and Employment Outcomes
Brief Title: Housing for Recovery Initiative
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Adrienne Sabety (Other)
Collaborators: Ohio Recovery Housing (Unknown); Ohio State University (Other)
Responsible Party: Sponsor-Investigator, Adrienne Sabety, Wilson Family LEO Assistant Professor of Economics, University of Notre Dame
Organization: University of Notre Dame (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-09-6787
Record Dates: First submitted 2022-02-24; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Substance-related Disorders; Alcohol-related Disorders; Housing
MeSH Terms: conditions — Substance-Related Disorders; Alcohol-Related Disorders

STUDY DESIGN:
Intervention Model Description: Study participants will be added to one of two arms, treatment (recovery housing) or control (no recovery housing), through a structured waitlist. If a placement in recovery housing becomes available for an individual within two weeks of when they are placed on the waitlist for housing, they will be in the treatment group. If a placement does not become available for an individual within two weeks of when they are added to the waitlist, they will be in the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recovery Housing (Experimental): Individuals in this arm will have access to a placement in recovery housing and the associated services. Recovery housing organizations provide individuals recovering from substance use disorders with housing and a variety of services, including transportation, rental assistance, life skills, family services, and educational and employment opportunities.
  Interventions: Behavioral: Recovery housing
- No Recovery Housing (No Intervention): Individuals in this arm will not receive a placement in recovery housing. When possible, they will be informed about other available services in their community.

INTERVENTIONS:
Behavioral: Recovery housing — Recovery housing provides housing and other services to individuals who are recovering from substance-use disorders. They provide a substance-free living environment, as well as services to assist residents with life in recovery. These services include connections to employment and educational opportunities, help obtaining documentation such as a driver's license, connection to mutual aid, and assistance building life skills.
  Arms: Recovery Housing

SUMMARY:
Recovery housing is a substance-free group home for those exiting drug and alcohol treatment. Individuals live in a recovery-focused environment with others traveling the same journey. Ohio Recovery Housing (ORH) creates and maintains standards of excellence for recovery housing in the state. Each house decides how it operates, with four different "levels" of housing available. These environments have the potential to help build a strong foundation in recovery to improve health, employment, and housing outcomes.

ORH and LEO will launch a quasi-experimental study to measure the impact of recovery housing for individuals with substance use disorders. The design relies on variation in the availability of program spots to identify effects. Invitations to join a home will come from a waitlist. As the length of the waitlist is unrelated to applicant characteristics, movement off the waitlist can be considered essentially random. The research team will compare those who receive services to those who do not.

The researchers hypothesize that those who participate in recovery housing will have improved health, employment, and housing outcomes compared to individuals who do not receive recovery housing services.

DETAILED DESCRIPTION:
The impact of ORH's recovery housing program will be evaluated using a quasi-experimental research design.

1. Individuals referred to or interested in recovery housing services typically contact an individual recovery home, either by phone or in person. At that time, ORH operator staff will screen individuals using existing eligibility criteria to determine if the individual would be a good fit for their recovery housing program. For example, clients must agree to follow house rules, live in a group environment, and be substance free. If they are unwilling to agree to these terms, they are not eligible for the program.
2. Interested clients will then complete an intake survey that collects basic demographic information about the client, some data about their history of substance use, and some economic data. This data is collected online using survey software, such as Qualtrics, so the data will be recorded electronically for all referred individuals. People that visit a home in person will be asked to fill out the survey on a tablet or computer. Those who call the home will answer these questions verbally over the phone, and the operator will complete the online survey on their behalf. The operator will explain the study to those who are deemed eligible for services and then obtain informed consent for study participation. If the operator is unable to answer individuals' questions, the operator will refer clients to the research team using the contact information provided on the informed consent form. For consenting individuals, identifying information will be collected for the purposes of tracking outcomes in administrative data and conducting a follow-up survey.
3. Eligible clients will be placed on a waitlist for the recovery housing program if there is not available capacity at the time they approach the program. If a program slot does not become available within two weeks, the individual will be removed from the waitlist and referred elsewhere. Individuals who are eligible for recovery housing based on the criteria set by ORH will have the same chance of receiving recovery housing services regardless of whether they consent to be in the study. All eligible individuals will be placed on the waitlist for housing in the order in which they arrive. Being part of the study will have no effect on an individual's ability to participate in recovery housing, and they will be clearly informed of this during the informed consent process.
4. Individuals for whom there is a recovery housing program slot available will be invited to move into the recovery home and receive specific provider services. All recovery housing providers in the ORH network will provide a healthy and safe environment, support for recovery planning, peer support services, referral to additional services in the community as identified by the resident's recovery plan, formal and informal recovery activities, and connection to mutual aid groups. Consenting individuals who are given a placement in recovery housing may choose to withdraw from the study at any point, including after they have been accepted into a recovery home. Withdrawing from the study will have no bearing on the services offered, nor the individual's relationship with ORH or affiliated providers.
5. Individuals for whom there is no program slot available will be assigned to the control group and will not have access to ORH recovery housing services. These individuals will be provided a list of other possible services elsewhere. Individuals placed in the control group will be able to re-enter the waitlist by contacting the recovery house to which they applied. Based on information provided by the recovery housing organizations, this will likely be a rare situation. For the purposes of analysis, individuals will be placed in the treatment or control group based on their assignment from the first time they are on the waitlist.
6. The research team will track outcomes of those who consented to be part of the study in administrative data sources to learn about housing stability, hospitalizations, and employment. These administrative records include inpatient stays and emergency department visits (collected by state Medicaid programs), earnings from employment as recorded by state unemployment insurance systems, and address histories from private address tracking services such as Infutor.
7. The data sharing agreements that would allow us to use these administrative data sources are in process. For example, LEO is currently working on data sharing agreements with the Ohio Department of Job and Family Services and the Ohio Department of Medicaid to obtain data on outcomes.
8. There are some key outcomes that cannot be derived from administrative sources. For example, sobriety among participants in the control group can only be quantified through an in-person survey. During the intake survey, personally identifiable information will be collected to perform a follow-up in-person survey.

ELIGIBILITY:
Inclusion Criteria:

* Individuals must have a history of, or a current problem with, substance abuse
* Individuals must be interested in starting or maintaining a lifestyle in which they do not use illicit drugs or drink alcohol
* Individuals must understand that recovery housing programs do not provide psychiatric services
* Individuals must be in recovery and prepared to live in a recovery housing environment

Exclusion Criteria:

* Individuals who are under the age of 18
* Individuals who do not consent to study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2430 (Estimated)
Dates: Start 2022-04-18 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Difference in maintenance of sobriety between treatment and control groups | 12 months after study enrollment
  Using survey data, we will quantify the effect of recovery housing participation on maintaining sobriety past 30 days and 6 months after the treatment group leaves housing. We will also measure the types of substances used (for example, alcohol, opioids,

SECONDARY OUTCOMES:
Differences in measures of personal relationships between treatment and control groups | 12 months after study enrollment
  We will use survey data to measure personal relationship outcomes, such as marital/cohabitation status and whether individuals have children in the custody of child welfare.
Differences in measured health and social insurance coverage between treatment and control groups | Up to 30 months after study enrollment
  We will use survey data to measure whether individuals have health insurance coverage other than Medicaid and whether they are enrolled in SNAP or TANF. We will use administrative data from the state of Ohio to measure Medicaid, SNAP, and TANF utilization.
Differences in criminal justice system involvement between treatment and control groups | Up to 30 months after study enrollment
  We will measure criminal justice outcomes by linking to publicly available criminal records, like county jail and state prison bookings records, as well as through survey data.
Differences in measures of housing stability between treatment and control groups | Up to 30 months after study enrollment
  We will use survey data to measure individuals' living arrangements (for example, in a house or apartment owned or leased in their own name, in a shared home or apartment, etc.) We will also ask retrospective questions about how many address changes they have had since exiting the waitlist. We will also measure housing stability with administrative data from Notre Dame's Infutor database.
Difference in measured health care access and utilization between treatment and control groups | Up to 30 months after study enrollment
  Using survey data, we will measure whether the respondent has a primary care provider, number of doctors' office visits, number of emergency department visits, number of prescription drug fills, and number of inpatient hospital stays in the previous six months. We will also survey individuals' self-reported physical and mental health status as well as a PHQ-2 screener for depression. We will also measure number of doctors' office visits, number of emergency department visits, number of prescription drug fills, and number of inpatient hospital stays in the previous six months using Ohio Medicaid data. We will use the Master Death Index to measure mortality.
Difference in measurement of employment and financial well-being between treatment and control groups | Up to 30 months after study enrollment
  We will use survey data to measure whether the individual has been employed over the last quarter, quarterly labor earnings, usual hours worked per week, and weeks worked over the past quarter. We also plan to use administrative data from the Ohio Department of Job and Family Services to collect data on whether the individual was employed in the last quarter and quarterly earnings. We will collect data on credit scores and use of credit from Experian.

CONTACTS AND LOCATIONS:
Overall Officials: Adrienne Sabety, PhD, Principal Investigator — University of Notre Dame; Mary Kate Batistich, PhD, Principal Investigator — University of Notre Dame; William Evans, PhD, Principal Investigator — University of Notre Dame; Thomas Gregoire, PhD, Principal Investigator — Ohio State University; Danielle Gray, MPH, Principal Investigator — Ohio Recovery Housing

IPD SHARING:
Plan to Share IPD: No